CLINICAL TRIAL: NCT04538001
Title: A Prospective, Multicenter, Randomized Trial in Evaluating the Safety and Efficacy of the Rotator Cuff Function Restoration Balloon in Patients With Irreparable Rotator Cuff Tear
Brief Title: Safety and Efficacy of Rotator Cuff Function Restoration Balloon in Irreparable Rotator Cuff Tear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHEER-I
Record Dates: First submitted 2020-08-14; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon implantation (Experimental): Arthroscopic implantation of this sub-acromial balloon
  Interventions: Device: Balloon implantation
- Rotator cuff repair (Active Comparator): Partial rotator cuff repair
  Interventions: Procedure: Rotator cuff repair

INTERVENTIONS:
Device: Balloon implantation — Subjects will undergo arthroscopic surgical intervention of debridement, long head of biceps tenotomy if deemed necessary with or without acromioplasty, and balloon implantation.
  Arms: Balloon implantation
Procedure: Rotator cuff repair — Subjects will undergo arthroscopic surgical intervention of debridement, long head of biceps tenotomy if deemed necessary with or without acromioplasty, and partial repair
  Arms: Rotator cuff repair

SUMMARY:
This study is a prospective, multicenter, randomized, controlled clinical study aiming to evaluate the safety and efficacy of the rotator cuff function restoration balloon in patients with irreparable rotator cuff tear compared to partial repair of the rotator cuff.

DETAILED DESCRIPTION:
This prospective, multicenter, randomized controlled clinical study is designed to enroll 112 subjects with irreparable rotator cuff tear and randomly assign them to the trial and control groups on a 1:1 basis.The experimental group was treated with rotator cuff restoration balloon, and the control group was treated with rotator cuff partial repair. The main end point of the study was improvement of the Constant Score at 6 months after the surgery. All subjects were followed up clinically at 1 day, 6 weeks, 3 months, 6 months and 1 year after the surgery, and were followed up with imaging examination at 3 months, 6 months and 1 year after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent pain and failure of non-operative treatment of the affected shoulder for at least 3 months
2. Failed non-operative treatment of at least 3 months
3. Patients are able to understand the purpose of the trial, voluntarily participated in and acknowledged the risks and benefits by signing the informed consent form
4. Patients can complete the clinical trial psychologically, physiologically and mentally, and can comply with all post-operative evaluations and visits
5. Posterosuperior rotator cuff tear diagnosed by MRI in the past 6 months, defined as the rotator cuff tear involving supraspinatus and infraspinatus muscles, and could be combined with type I subscapular muscle injury.
6. Evidence of any one of the following conditions confirmed by MRI:

(1) The rotator cuff tear measuring >3cm in size; (2) involving ≥ 2 tendons; (3) stage 3 or 4 fatty infiltration according to Goutallier Classification; (4) acromiohumeral interval <7mm. 7. All subjects meeting the above inclusion criteria will undergo arthroscopic debridement, if the tear size is still >3cm at medial to lateral direction, and the superior edge cannot be fixed to the footprint area to overlap bone coverage for complete repair.

Exclusion Criteria:

1. Known allergy to the balloon material (polyethylene)
2. Evidence of osteoarthritis or cartilage damage in the shoulder
3. Evidence of gleno-humeral instability or axillary nerve palsy
4. Evidence of major joint trauma, infection, or necrosis in the shoulder
5. Previous surgery of the index shoulder in the past 1 year, excluding diagnostic arthroscopy
6. Shoulder pain due to other unknown causes
7. Major medical condition or known drug or alcohol abuses that could affect quality of life and influence the results of the study.
8. Subjects with poor compliance, unable to complete the trial according to the requirements or for other reasons, or considered not to be suitable for inclusion by investigators.
9. Concurrent participation in any other invasive clinical study one month prior to enrollment to the study and during the entire study period.
10. Acute infection requiring antibiotics
11. Subjects receiving prescription narcotic pain medication for conditions unrelated to the index shoulder condition
12. Subjects with implanted metallic devices (e.g., cardiac pacemakers, insulin pumps, nerve stimulators) or other contraindications for MRI scan
13. Severe dysfunction in heart, brain, lungs or kidney and cannot tolerate surgery.
14. Severe disorder in bleeding or coagulation function that cannot be corrected.
15. Pregnancy
16. Subjects being suffered from other serious illness which may affect quality of life the results of the study (e.g. HIV, active malignancy in the past 5 years, transmural myocardial infarction in 6 months, unstable angina pectoris, CVA, renal insufficiency, etc.)
17. Diseases or other conditions which cannot finish 1 year follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Constant-Murley shoulder outcome score | 6 months post operation
  Change in Constant-Murley shoulder outcome score and improvement compare to baseline

SECONDARY OUTCOMES:
Change in Constant-Murley shoulder outcome score | 3 months, 1year post operation
  Change in Constant-Murley shoulder outcome score and improvement compare to baseline at each time point
Change in American Shoulder and Elbow Score (ASES) | 3 months, 6 months and 1year post operation
  Change in American Shoulder and Elbow Score (ASES) and improvement compare to baseline at each time point
Change in pain score | 1 day, 6weeks, 3 months, 6months, 1year post operation
  Change in Visual Analog Scale pain score and improvement compare to baseline at each time point
Change in range of motion | 3 months, 6months, 1year post operation
  Change in range of motion and improvement compare to baseline at each time point, including active shoulder flexion and extension (from ASES score)
Acromiohumeral distance | 3 months, 6months, 1year post operation
  The distance between the acromion and the proximal humerus
Safety assessment | Peri-operation and 1 day, 6weeks, 3 months, 6months, 1year post operation
  The Safety assessment will include the incidence of AEs/SAEs throughout the entire study period

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices) will be shared. Additionally, study protocol will be available. The data will become available for the beginning 3 months and ending 5 years following article publication. The access criteria are as follow:
  (With) Researchers who provide a methodologically sound proposal. (For the analysis) to achieve aims in the approved proposal. (Requisite mechanism) Proposals should be directed to mzheng@microport.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).
  If the data sharing plan changes after registration, this should be reflected in the statement submitted and published with the manuscript, and updated in the registry record.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: * (With) Researchers who provide a methodologically sound proposal.
  * (For the analysis) to achieve aims in the approved proposal.
  * (Requisite mechanism) Proposals should be directed to mzheng@microport.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).